CLINICAL TRIAL: NCT02342444
Title: A Prospective Randomized Trial Comparing Two Standard Doses of Enoxaparin for the Prevention of Thromboembolism in Surgical Patients
Brief Title: Lovenox 30 mg Twice Daily (BID) Versus 40 mg Once Daily (QD)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Martin A Schreiber, MD, Professor & Chief of Trauma, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8080
Record Dates: First submitted 2014-05-21; First posted 2015-01-21 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Trauma; Surgery; Deep Vein Thrombosis (DVT); Thromboembolic Events
Keywords: Trauma; Surgery; Enoxaparin; DVTs; Thromboembolic events
MeSH Terms: conditions — Wounds and Injuries; Venous Thrombosis; Thromboembolism | interventions — enoxaparin sodium; BID protein, human; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enoxaparin Sodium Injection 30 mg BID (Active Comparator): Subjects are randomized to receive 30 mg twice daily of enoxaparin.
  Interventions: Drug: Enoxaparin Sodium Injection 30 mg BID
- Enoxaparin Sodium Injection 40 mg QD (Active Comparator): Subjects are randomized to receive 40 mg once daily of enoxaparin.
  Interventions: Drug: Enoxaparin Sodium Injection 40 mg QD

INTERVENTIONS:
Drug: Enoxaparin Sodium Injection 30 mg BID
  Other Names: Lovenox
  Arms: Enoxaparin Sodium Injection 30 mg BID
Drug: Enoxaparin Sodium Injection 40 mg QD
  Other Names: Lovenox
  Arms: Enoxaparin Sodium Injection 40 mg QD

SUMMARY:
The risk of developing a blood clot occurs in up to 60% of all critical care patients. Many times enoxaparin (or Lovenox) is given to patients who are at a higher risk of developing clots in their legs or lungs. There are two standard doses of enoxaparin that are recommended by the drug companies. These two doses have never been directly compared in trauma, general, and vascular surgery patients. The purposes of this study are:

1. to compare the development of blood clots in patients receiving 30mg twice daily of enoxaparin compared to patients receiving 40mg once daily of enoxaparin.
2. to determine if there is higher risk of bleeding complications in patients receiving 30mg twice daily of enoxaparin compared to patients receiving 40mg once daily.

Patients enrolled into the study will be randomized to receive enoxaparin, 30mg twice daily or enoxaparin, 40mg once daily. Patients will then be monitored for signs and symptoms of blood clots. At the time of discharge (or before, if medically indicated), an ultrasound test will be performed to look for blood clots in the patient's legs.

The investigators will compare incidence of blood clots formed between the 2 groups of patients to determine if one dose of enoxaparin relates to a lower rate of blood clots in critically ill patients. The investigators will also compare the incidence of bleeding complications between the 2 groups.

DETAILED DESCRIPTION:
This is a prospective randomized single center study in human subjects.

Initiation of enoxaparin thromboprophylaxis will be done by the treatment team. Patients admitted to the trauma service will be eligible for enrollment. Research staff will approach patients or their LARs for consent prior to or at the time enoxaparin is ordered. This will include patients with traumatic intracranial hemorrhage, after the consulting neurosurgical team and primary treatment team decide to initiate thromboprophylaxis. Once enrolled, the subject will be randomized to receive either 30 mg twice daily dosing or 40 mg daily dosing of enoxaparin. However, treatment team will be responsible for deciding when to start enoxaparin treatment. Patients who are discharged without receiving enoxaparin or are started on a non-standard or therapeutic dose will be withdrawn from the study. Patient characteristics: age, sex, body mass index (BMI), medical comorbidities, Acute Physiology and Chronic Health Evaluation II score (APACHE II), injuries, and operations will be collected, coded with a unique identification letter and number combination, and entered into a database.

All patients will undergo weekly ultrasound duplex examination of the lower extremities for the presence of deep venous thrombosis. Patients who develop symptoms of pulmonary embolism including acute shortness of breath and increased A-a gradient will undergo computed tomography angiography as part of their standard care. A bleeding complication will be defined as a known bleeding episode associated with hypotension (greater than 20 mmHG drop from baseline) and the need for blood transfusion.

Current practice at OHSU is for patients age 15 and above to be admitted to the adult trauma service, and are treated with the same standard of care as adults. Currently, there are no clear data stratifying the risk of VTE in this population compared to other age groups. Therefore, patients in this age range on the adult Trauma Service will be included in the study as they are treated in the same method as our adult patient population.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients requiring prophylactic dosing of enoxaparin (Lovenox)
* Admitted to the trauma or surgical service
* Age greater than 15 years

Exclusion Criteria:

* Unable to obtain consent from patient or authorized representative
* Presence of intracranial hemorrhage
* Receiving therapeutic dose of enoxaparin (Lovenox)
* Receiving other forms of anticoagulation
* Presence of renal failure requiring non-standard dosing regimen

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic events | Daily, up to Day 90
  Daily monitoring per standard of care for the development of thromboembolic events.

SECONDARY OUTCOMES:
Increase in bleeding complications | Daily, up to Day 90
  Daily monitoring for an increase in bleeding complications due to study drug dose and regime.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Schreiber, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States